CLINICAL TRIAL: NCT04353726
Title: Individualized Diet Improvement Program (iDip) for Weight Loss and Maintenance.
Brief Title: Knowledge-based Dietary Weight Management.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Mindy Lee, Graduate Research Assistant, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18069
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Weight Loss; Dietary Modifications; Obesity; Sustainability
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Intervention Model Description: Before and after study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Eligible participants will be in an intervention group led by a registered dietitian
  Interventions: Other: Weight management

INTERVENTIONS:
Other: Weight management — During a 12-month period, participants will attend a total of 22 diet improvement sessions, each of which will last approximately 1 hour. Twelve sessions will be held in the first 5 months and will be focused on safe and efficient weight loss. The participants will learn to create a personalized weight loss diet from their kitchen based on their diet practice and food preference. The next 10 sessions will be held in the last 7 months and will be focused on weight maintenance and healthy eating. The participants will build skills to select foods and create meals that prevent them from overeating.

SUMMARY:
This research is to develop a weight loss and weight maintenance program through dietary modifications for adults with obesity. Although scientific studies have shown the feasibility of rapid and safe dietary weight loss and subsequent weight maintenance, no efficacious dietary weight management program is widely available, and thus bariatric surgery remains the most reliable approach for weight loss/management. Safe and effective dietary weight loss and subsequent weight maintenance require flexible, individualized advice by an experienced dietitian/nutritionist.

ELIGIBILITY:
Inclusion criteria:

* age 18-64 years;
* body mass index (BMI) >28 kg/m2;
* not currently pregnant or lactating;
* have Wi-Fi at home, a working email, and an iPhone or Android smartphone.
* no self-reported severe metabolic, cardiovascular or musculoskeletal disease;
* not using insulin injection;
* able to attend the 22 (1 hour) diet improvement sessions.
* willing to lose 20 lb. or more for 6 months and maintain a healthy weight for one year.
* keep weighing their weight for one and a half years.
* fluent in reading and writing English.

Exclusion criteria:

* age <18 or >64 years;
* body mass index of <28 kg/m2;
* currently pregnant;
* currently lactating;
* self-reported with the severe metabolic, cardiovascular or musculoskeletal disease;
* use insulin injection;
* not able to attend the 22 (1 hour) diet improvement sessions for 1 year;
* failed to set up a Wi-Fi scale;
* failed to submit a food frequency questionnaire

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Body weight | Change from baseline body weight at 6 months
  Body weight in kilograms
Body weight | Change from baseline body weight at 12 months
  Body weight in kilograms
Body weight | Change from baseline body weight at 18 months
  Body weight in kilograms

SECONDARY OUTCOMES:
Waist circumference | Change from baseline waist circumference at 12 months
  Waist circumference in centimeters
Hip circumference | Change from baseline hip circumference at 12 months
  Hip circumference in centimeters
Protein intake | Change from baseline protein intake at 6 months
  Protein intake in grams and caloric intake will be combined to report density in g/100kcal
Protein intake | Change from baseline protein intake at 12 months
  Protein intake in grams and caloric intake will be combined to report density in g/100kcal
Fiber intake | Change from baseline fiber intake at 6 months
  Fiber intake in grams and caloric intake will be combined to report density in g/100kcal
Fiber intake | Change from baseline fiber intake at 12 months
  Fiber intake in grams and caloric intake will be combined to report density in g/100kcal

CONTACTS AND LOCATIONS:
Overall Officials: Nakamura T Manabu, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be maintained for three years after completion of the study
Access Criteria: Findings will be disseminated via abstracts and presentations at scientific conferences and through manuscripts and journal articles within the field.